CLINICAL TRIAL: NCT00926237
Title: Effect of rTMS on Resting State Brain Activity in Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 109033
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Tinnitus
Keywords: Tinnitus; Transcranial Magnetic Stimulation; TMS; rTMS
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham followed by active 1Hz, then active 10Hz rTMS (Experimental): Subjects assigned to this arm received sham rTMS followed by active rTMS at 1Hz and then active rTMS at 10 Hz. Each treatment consisted of a four-day trial with no less than 21 days separating each condition. Subjects receive sham stimulation first to prevent carry forward effects of the active treatment condition into the sham condition.
  Interventions: Device: Sham rTMS - Sham repetitive transcranial magnetic stimulation; Device: Active 1 Hz rTMS - Active repetitive transcranial magnetic stimulation delivered at 1 Hz frequency; Device: Active 10 Hz rTMS - active repetitive transcranial magnetic stimulation delivered at 10 Hz frequency
- Sham followed by active 10Hz and active 1Hz rTMS (Experimental): Subjects assigned to this arm received sham rTMS followed by active rTMS at 10 Hz and then active rTMS at 1 Hz. Each treatment consisted of a four-day trial with no less than 21 days separating each condition. Subjects receive sham stimulation first to prevent carry forward effects of the active treatment condition into the sham condition.
  Interventions: Device: Sham rTMS - Sham repetitive transcranial magnetic stimulation; Device: Active 1 Hz rTMS - Active repetitive transcranial magnetic stimulation delivered at 1 Hz frequency; Device: Active 10 Hz rTMS - active repetitive transcranial magnetic stimulation delivered at 10 Hz frequency

INTERVENTIONS:
Device: Sham rTMS - Sham repetitive transcranial magnetic stimulation — Sham rTMS will be delivered using a commercially available sham coil and targeted to the same brain site in the temporal lobe and in a manner identical to that for active rTMS except that scalp electrodes are used to stimulate the temporalis muscle electrically during sham stimulation to replicate the feel of active TMS.
Device: Active 1 Hz rTMS - Active repetitive transcranial magnetic stimulation delivered at 1 Hz frequency — Active rTMS will be targeted either to the mid-superior temporal gyrus opposite the ear with loudest tinnitus or to the same region in the left hemisphere if no asymmetry in tinnitus is present. 1 Hz active rTMS will be delivered at 110% of motor threshold (MT) for a total of 1800 magnetic pulses per session, 4 sessions per week.
Device: Active 10 Hz rTMS - active repetitive transcranial magnetic stimulation delivered at 10 Hz frequency — Active rTMS will be targeted either to the mid-superior temporal gyrus opposite the ear with loudest tinnitus or to the same region in the left hemisphere if no asymmetry in tinnitus is present. 10 Hz active rTMS will be delivered at 110% of motor threshold (MT) for a total of 1800 magnetic pulses per session, 4 sessions per week.

SUMMARY:
One out of every five people experiences tinnitus (a ringing, buzzing, or roaring sound in the ear) ranging from mild to severe impairment. To date, there are no effective therapies available that have been shown to decrease tinnitus awareness. The purpose of this study is to evaluate a treatment option for tinnitus that uses a technique called Repetitive Transcranial Magnetic Stimulation (rTMS), which could prove to be an effective means of alleviating or reducing the symptoms of tinnitus.

DETAILED DESCRIPTION:
Up to 60 subjects, including males and females ages 19-89 years old and of all races, and with tinnitus severe enough to seek medical attention, will be enrolled in this study. All participants must be evaluated or have documentation of being evaluated prior to beginning therapy with rTMS in order to confirm eligibility and to rule out any medically treatable causes of tinnitus. An MRI scan of the head may or may not be required, depending upon the results of this evaluation, in order to rule out specific middle ear pathologies.

This study will require participation in at least three weeks (4 weekdays per week) of rTMS sessions, including two active weeks and a sham (or placebo) week. There will be a three week washout period following each treatment week. At the completion of the three treatment weeks, subjects who have noticed an improvement in their tinnitus will have the option of participating in a maintenance rTMS program providing up to 8 additional weeks of treatment.

ELIGIBILITY:
Inclusion Criteria per protocol and informed consent:

* Diagnosis of tinnitus established through a history and physical exam or review of records.
* Subjects 19-89 years of age
* Tinnitus present for at least 6 months and severe enough to seek medical attention
* Subjects taking SSRI's (a class of anti-depressant medications)and benzodiazepines (a class of anti-anxiety medications) for depression or anxiety related to tinnitus must be stable on their current dose for at least 3 months and must not alter their dose or medication during their involvement with this study
* Subjects must agree to avoid consuming alcohol within 72 hours of each rTMS session
* Female subjects of childbearing potential must demonstrate a negative pregnancy test during their initial clinic visit and must agree to use effective contraception during their participation in this study
* Subjects must sign an informed consent and agree to comply with study and follow-up procedures, including completion of all necessary questionnaires and testing, as well as, being video-recorded for safety purposes during rTMS sessions
* Subjects must speak and comprehend English adequately to understand and complete any study-related instructions and questionnaires

Exclusion Criteria per protocol and informed consent:

For rTMS

* Subjects or any of their 1st-degree relatives must not have been diagnosed with epilepsy
* Subjects must not have a history of seizure disorder or migraines
* Subjects must not have any history of a brain aneurysm, stroke, previous cranial neurosurgery, acoustic neuroma, glomus tumor, active Menniere's Disease, profound hearing loss (greater than 90 dB at 4000 Hz), or any major neurological or psychiatric disorders (excluding depression or anxiety related to tinnitus)
* Medications that lower seizure threshold or reduce cortical excitation (i.e., tricyclic antidepressants, bupropion or anticonvulsants)
* Subjects must not have any history of a head injury that resulted in a loss of consciousness for more than 10 minutes
* Subjects must not be pregnant or refuse to utilize effective contraception during their participation in this study For MRI
* Subjects must not have any metal implants or devices in the head or neck or a pacemaker.
* Subjects must not have severe claustrophobia if they are to have an MRI.
* Significant abnormalities must not be present on acquired or existing CT or MRI image of the head.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mennemeier, PhD, Principal Investigator — UAMS Department of Neurosciences
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 58 participants were enrolled. Recruitment used a waitlist of subjects who already expressed interest in tinnitus studies and from advertisement.
Pre-assignment Details: Of the 58 subjects enrolled, only 39 were assigned to study groups. Two subjects who initially failed screening were re-enrolled via a waiver before assignment. Ten had participated in an early version of the protocol that was not comparable. Seven subjects dropped out after baseline. So 2+10+7= the 19 participants who were enrolled but not started in the participant flow.
Groups:
- Sham Followed by Active 1Hz Then 10Hz rTMS: Subjects assigned to this arm received sham rTMS followed by active rTMS at 1Hz and then active rTMS at 10 Hz. Each treatment consisted of a four-day trial with no less than 21 days separating each condition. Subjects receive sham stimulation first to prevent carry forward effects of the active treatment condition into the sham condition.
  Sham rTMS
  Active 1 Hz rTMS
  Active 1 Hz rTMS
- Sham Followed by Active 10Hz Then 1Hz rTMS: Subjects assigned to this arm received sham rTMS followed by active rTMS at 10 Hz and then active rTMS at 1 Hz. Each treatment consisted of a four-day trial with no less than 21 days separating each condition. Subjects receive sham stimulation first to prevent carry forward effects of the active treatment condition into the sham condition.
  Sham rTMS
  Active 1 Hz rTMS
  Active 10 Hz rTMS
Period: Overall Study
Arm/Group | Sham Followed by Active 1Hz Then 10Hz rTMS | Sham Followed by Active 10Hz Then 1Hz rTMS
Started | 19 (Two subjects withdrew after receiving sham rTMS but before receiving active rTMS.) | 20 (One subjects withdrew after receiving sham rTMS but before receiving active rTMS.)
Completed | 17 | 19
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Numbers are reported for all persons enrolled in the study, not just those for subjects who were assigned to a treatment arm.
Groups:
- All Subjects Enrolled in the Study: Baseline information is reported for all subjects enrolled.
Arm/Group | All Subjects Enrolled in the Study
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 56
  More than one race | 1
  Unknown or Not Reported | 0
Baseline analogue ratings of tinnitus awareness [Mean (Standard Deviation); unit: units on a scale] — Baseline ratings are the average of the baseline assessments on separate days. Analogue ratings of tinnitus awareness range from 0 (no tinnitus) to 100 (painfully loud tinnitus). Population: Baseline ratings are reported only for the 39 subjects who were assigned to a treatment arm and completed all baseline assessments
  units on a scale
    number analyzed (Participants) | 39
    (all) | 58.72 (22.56)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Analogue Rating of Tinnitus Awareness.
Description: Change from baseline on the daily analogue rating of tinnitus awareness. Analogue ratings are a validated self report instrument assessing subjects awareness of tinnitus in daily life. Possible scores range from 0 (no tinnitus) to 100 (painfully loud tinnitus). Change equals the average rating for a given treatment week or washout period minus the average rating over three baseline assessments.
Time Frame: from baseline to: day 6 (sham), day 25 (sham w/o), day 29 (1st active TX), day 50 (1st active w/o), day 50 (2nd active TX), day 76 (2nd active w/o).
Population: The analysis population includes 36 subjects who completed the all baseline, sham rTMS, sham washout, active 1 Hz rTMS, 1Hz washout, active 10Hz rTMS and 10Hz washout periods.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Sham rTMS: This comparison examined change in analogue ratings of tinnitus awareness between the baseline and the sham rTMS treatment condition.
- Sham Washout: This comparison examined change in analogue ratings of tinnitus awareness between baseline and the sham washout period of 21 days.
- 1 Hz Active rTMS: This comparison examined change in analogue ratings of tinnitus awareness between the baseline and the 1 Hz active rTMS condition.
- 1 Hz Washout: This comparison examined change in analogue ratings of tinnitus awareness between baseline and the 1 Hz washout period lasting 21 days.
- 10 Hz Active rTMS: This comparison examined change in analogue ratings of tinnitus awareness between the baseline and the 10 Hz active rTMS condition.
- 10 Hz Washout: This comparison examined change in analogue ratings of tinnitus awareness between baseline and the 10 Hz washout period of 21 days.
Arm/Group | Sham rTMS | Sham Washout | 1 Hz Active rTMS | 1 Hz Washout | 10 Hz Active rTMS | 10 Hz Washout
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36
units on a scale | -4.08 (3.72) | -4.70 (3.90) | -9.82 (3.72) | -9.89 (3.91) | -10.85 (3.85) | -9.43 (4.06)
Statistical Analysis 1: Comparison: Sham rTMS vs 1 Hz Active rTMS; Test type: Superiority; p = .04, Mixed Models Analysis — t value = -1.40; Mean Difference (Final Values) = -5.74 — 1Hz active rTMS - Sham rTMS
Statistical Analysis 2: Comparison: Sham rTMS vs 10 Hz Active rTMS; Test type: Superiority; p = .02, Mixed Models Analysis — t value = -2.03; Mean Difference (Final Values) = -6.77 — 10 Hz active rTMS - Sham rTMS
Statistical Analysis 3: Comparison: Sham Washout vs 10 Hz Washout; Test type: Superiority; p = .20, Mixed Models Analysis — t value = -1..28; Mean Difference (Final Values) = -4.73 — 10 Hz washout - sham washout period
Statistical Analysis 4: Comparison: Sham Washout vs 1 Hz Washout; Test type: Superiority; p = .19, Mixed Models Analysis — t value = -1.29; Mean Difference (Final Values) = -5.19 — 1Hz washout - sham washout

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline until study completion at followup: ~113 days for participants who did not enter maintenance and up to ~159 days for subjects who entered maintenance.
Description: While it was possible to accurately report Adverse Events by assigned Arm, it was not possible to accurately report adverse events by rTMS frequency because the majority of adverse events (49/58) were not study related. Rather they included illness or injuries that occurred outside the study in daily life. Only 9/58 adverse events were coded as study related and these are described in the Adverse Event Additional Description field.
Groups:
- Subjects Who Received Sham Followed by Active 1 Hz rTMS Then Active 10 Hz rTMS.: Subjects in this arm received a course of sham stimulation which was followed by a course of active stimulation at 1 Hz rTMS and then a course of active stimulation at 10 Hz.
- Subjects Who Received Sham Followed by Active 10 Hz rTMS Then Active 1 Hz rTMS: Subjects in this arm received a course of sham stimulation which was followed by a course of active stimulation at 10 Hz rTMS and then a course of active stimulation at 1 Hz.
Arm/Group | Subjects Who Received Sham Followed by Active 1 Hz rTMS Then Active 10 Hz rTMS. | Subjects Who Received Sham Followed by Active 10 Hz rTMS Then Active 1 Hz rTMS
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/31
Other Adverse Events (participants affected / at risk) | 12/27 | 8/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Who Received Sham Followed by Active 1 Hz rTMS Then Active 10 Hz rTMS. (N=27) | Subjects Who Received Sham Followed by Active 10 Hz rTMS Then Active 1 Hz rTMS (N=31)
Death (Cardiac disorders) | 1 | 0 — Drowning. Not study related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Who Received Sham Followed by Active 1 Hz rTMS Then Active 10 Hz rTMS. (N=27) | Subjects Who Received Sham Followed by Active 10 Hz rTMS Then Active 1 Hz rTMS (N=31)
Headache (Skin and subcutaneous tissue disorders) | 4 | 4 — In the 1 Hz first arm 4/4 reports of headache were coded as related to the study intervention; whereas in the 10 Hz first arm 1/4 reports of headache were study related.
Jaw pain (Musculoskeletal and connective tissue disorders) | 3 | 1 — In the 1 Hz first arm 3/3 reports of jaw pain were coded as related to the study intervention; whereas in the 10 Hz first arm 0/1 reports were study related.
Tinnitus increase (Nervous system disorders) | 1 | 0 — In the 1 Hz first arm 1/1 reports of tinnitus increase were coded as related to the study intervention; whereas in the 10 Hz first arm there were no such reports.
Illness (General disorders) | 11 | 7 — reported illness not due to intervention (Flu, orthopedic, back pain, injury)
eye muscle twitching (Eye disorders) | 0 | 2 — report of eye muscles twitching after intevention
Increase heart rate (Cardiac disorders) | 1 | 0 — Report of increase heart rate prior to session.

LIMITATIONS AND CAVEATS:
Limited recruitment and retention into maintenance (n=3 with complete data) precluded meaningful data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT00926237/Prot_SAP_000.pdf